CLINICAL TRIAL: NCT03813537
Title: Evaluation of Hospital Readmission Rate Dependent on Post-Operative Follow-Up Procedure: A Randomized Prospective Clinical Trial
Brief Title: Evaluation of Hospital Readmission Rate Dependent on Post-Operative Follow-Up Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syed Husain (Other)
Responsible Party: Sponsor-Investigator, Syed Husain, Assistant Professor - Colon and Rectal Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018H0207
Record Dates: First submitted 2018-05-24; First posted 2019-01-23 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to two arms:
  1. Intervention: post operative phone call with protocol driven follow up pathway.
  2. Control: Current standard post operative follow up practice at our institution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The control will be discharged with standard of care follow-up instructions and scheduled for a standard follow-up clinic visit within 2-3 weeks post-op.
- Phone Call (Experimental): The experimental group will receive a phone call intervention 3 days post-op. During this phone call, the patient will be asked questions using a study questionnaire based on the most frequent indications for readmission post colorectal surgery. Based on the responses, patients will be advised to maintain the scheduled appointment, visit the clinic within 48 hours, or go to the Emergency Department immediately.
  Interventions: Other: Phone Call

INTERVENTIONS:
Other: Phone Call — The experimental group will receive a phone call 3-days post procedure and asked questions based on the most frequent indications for readmission after colorectal surgery.
  Arms: Phone Call

SUMMARY:
This study is a randomized clinical trial among colorectal surgery patients that will compare the efficacy of two different discharge protocols - current standard of care follow-up at two weeks post-op versus a 3-day phone call intervention. The overall aim of the study is to identify areas of improvement for discharging and following patients within 30 days of colorectal surgery.

DETAILED DESCRIPTION:
This study will be a prospective clinical trial, in which colorectal surgery patients will be randomly assigned to a control or experimental group. Patients will be consented and randomized prior to discharge.The control group will be discharged with standard of care follow-up instructions described by The Ohio State University Wexner Medical Center (OSUWMC), and scheduled to come in for a standard follow-up clinic visit within 2-3 weeks. The experimental group will also be scheduled for a 2-3 week post-op follow-up appointment, but will also receive a phone call 3-days post procedure. During this phone call, the patient will be asked questions using a study-specific questionnaire that is based on the most frequent indications for readmission after colorectal surgery. Based on the responses, patients will be advised to maintain the scheduled 2-3 week post-op appointment, visit the clinic within 48 hours, or go to the Emergency Department immediately. To determine if patients had visited an ED or been readmitted to a hospital within 30 days of colorectal surgery, both the standard of care and intervention groups will receive a phone call 30-days post-discharge. At this time we will also conduct the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey to measure patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Patients who underwent colorectal surgery at The Ohio State University Wexner Medical Center

Exclusion Criteria:

* Patients under 18 years old
* Patients with limited ability to communicate
* Patients who do not have a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Post-Operative Phone Call (assess readmission rates) | 3 days
  Assess readmission rates

SECONDARY OUTCOMES:
Post Discharge Survey (assess patient satisfaction) | 30 days
  Assess patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Syed Husain, MBBS, Principal Investigator — OSU Wexner Medical Center
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No